CLINICAL TRIAL: NCT00540137
Title: A Randomised Prospective Study Assessing Changes in Neurocognitive Function, Using a Computerised Test Battery, in Treatment Naïve HIV-1 Positive Subjects Commencing Two Different Antiretroviral Regimens
Brief Title: The CogNaive Study: Assessing Changes in Neurocognitive Function in Treatment Naïve HIV-1 Positive Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudra-CT 2007-002405-47
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2010-05

CONDITIONS: HIV Infections
Keywords: Antiretroviral therapy; Neurocognitive function; Magnetic resonance spectroscopy; HIV disease; Treatment Naive
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nevirapine; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NRTIs plus NNRTI arm (Active Comparator): nevirapine 400 mg once daily (after 12 weeks induction)with a nucleoside backbone
  Interventions: Drug: nevirapine
- NRTIs plus PI arm (Active Comparator): atazanavir 300 mg once daily, ritonavir 100 mg once daily with a nucleoside backbone
  Interventions: Drug: atazanavir/ritonavir

INTERVENTIONS:
Drug: nevirapine — 400mg once daily
  Arms: NRTIs plus NNRTI arm
Drug: atazanavir/ritonavir — atazanavir 300 mg once daily ritonavir 100 mg once daily
  Arms: NRTIs plus PI arm

SUMMARY:
The purpose of this study is to investigate the possibility of an association between changes in neurocognitive function, as measured by a computerised test battery, and the use of two different highly active antiretroviral therapy (HAART) regimens in treatment naïve HIV-1 infected subjects commencing antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females
* Signed informed consent
* No previous antiretroviral treatment
* Males with CD4+ lymphocyte count < 400 cells/ųL and females with CD4+ lymphocyte count < 250 cells/ųL
* Susceptible to all currently licensed nucleoside reverse transcriptase inhibitors (NRTIs), non-nucleoside reverse transcriptase inhibitors (NNRTIs) and protease inhibitors (PIs)

Exclusion Criteria:

* Existing neurological disease
* Hepatitis B or hepatitis C co-infection
* Current history of major depression or psychosis
* Recent head injury
* Current alcohol abuse or drug dependence
* Active opportunistic infection or significant co-morbidities

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess changes in simple reaction time as measured by a computerised test battery | over study period

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Heart of England NHS Foundation Trust, Birmingham
  - St. Mary's Hospital, London